CLINICAL TRIAL: NCT00590421
Title: Carotid Atherosclerotic Disease Following Childhood Scalp Irradiation
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Shai Efrati, Assaf-Harofeh Medical Center
Other Study IDs: Car&RAD05; 57/04
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-12

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples, 10 ml, were procured for assessment of creatinine, total cholesterol, high density lipoproteins (HDL), triglycerides (TG), calculated low density lipoproteins (LDL) and homocysteine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 145 individuals treated by irradiation in their childhood
- 2: 150 matched control subjects with no history of irradiation

SUMMARY:
Background: During the first half of the 20th century, scalp irradiation was a standard treatment for induction of epilation in children suffering from Tinea Capitis. These children are now more than 50 years old and the aim was to investigate the possible association between their childhood low dose irradiation exposure and development of carotid atherosclerotic disease in adulthood.

Methods: The study included 145 individuals treated by irradiation in their childhood, and 150 matched control subjects with no history of irradiation. B-mode ultrasound imaging and US Doppler were used to measure carotid and femoral stenosis and Intima-Media Thickness (IMT). Blood samples were taken for lipid profile and homocysteine evaluation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* childhood scalp irradiation or mach controls
* writen informed consent

Exclusion Criteria:

* inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was designed to include 150 persons who were treated as children for Tinea Capitis by scalp irradiation in the 1950's and 150 subjects who were not exposed to radiation. This sample size was determined under the following assumption: power of ≥95%, alpha error level of 5%, 10% prevalence of carotid stenosis in the non exposed group and minimal OR of 2.5.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2004-07; Primary Completion 2007-01 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel